CLINICAL TRIAL: NCT05994014
Title: PET/CT vs. Cardiac CT for Detecting Coronary Atherosclerotic Disease
Brief Title: PET/CT* vs. Cardiac CT for Detecting Coronary Atherosclerotic Disease [*PET: Positron Emission Tomography; CT: Computed Tomography]
Acronym: PET; CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00317553
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Coronary Atherosclerosis of Native Coronary Artery
Keywords: coronary imaging; prevention; early detection
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Main group (Other): All patients undergo both, experimental and standard, tests
  Interventions: Diagnostic Test: PET/CT

INTERVENTIONS:
Diagnostic Test: PET/CT — Experimental test for detecting atherosclerosis

SUMMARY:
Early detection of coronary atherosclerotic disease facilitates adequate prevention. The purpose of this study is to compare an assessment of coronary atherosclerotic disease burden by positron emission tomography / computed tomography (NaF-PET/CT) with those of conventional and ultra-high-resolution-CT (UHR-CT) in patients with suspected coronary artery disease. For this purpose, the investigators plan to include 33 patients with symptoms concerning for CAD who have been referred for cardiac CT testing.

DETAILED DESCRIPTION:
Early detection of coronary atherosclerotic disease facilitates adequate prevention. 18 Fluoride (F) -sodium fluoride PET/CT (NaF-PET/ CT) has been shown to detect aortic microcalcification as early manifestation of atherosclerosis in experimental and early clinical investigations. The capability of NaF-PET/CT to detect coronary atherosclerotic disease in humans remains unclear. Given its sensitivity to detect vascular microcalcification undetectable by conventional CT, NaF-PET/CT may be an attractive, noninvasive test for early detection of coronary atherosclerosis.

The purpose of this study is to compare an assessment of coronary atherosclerotic disease burden by positron emission tomography / computed tomography (NaF-PET/CT) with those of conventional and ultra-high-resolution-CT (UHR-CT) in patients with suspected coronary artery disease (CAD). For this purpose, the investigators plan to include 33 patients with symptoms concerning for CAD who have been referred for cardiac CT testing. In addition to the clinically indicated and performed cardiac CT scan, participants will be asked to also undergo NaF-PET/CT for comparison of atherosclerosis assessment among the two tests (single center, prospective diagnostic accuracy study).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* 18 years or older
* referred for coronary CT angiography because of suspected coronary heart disease (CHD) with stable symptoms

Exclusion Criteria:

* The patient has a history of coronary heart disease, defined by prior myocardial infarction or prior coronary artery revascularization.
* Pregnancy.
* Atrial fibrillation.
* Morbid obesity defines as a body mass index of >40.
* The patient has any other clinically significant medical condition that in the opinion of the Investigator could impact the patient's ability to successfully complete the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Correlation of atheroma volume [mm3] | 60 days
  Coronary atheroma volume by PET/CT vs. CT total atheroma volume
Diagnostic accuracy of detecting coronary atherosclerosis | 60 days
  PET/CT Sensitivity to detect any atherosclerosis by CT angiography

CONTACTS AND LOCATIONS:
Overall Officials: Armin Zadeh, MD PhD MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States